CLINICAL TRIAL: NCT03565926
Title: Effects of Hipopressive Exercises Versus Manual Therapy in Subjects With Nonspecific Low Back Pain
Brief Title: Effects of Hipopressive Exercises in Nonspecific Low Back Pain
Acronym: HPvsMT-LBP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Valencia (Other)
Responsible Party: Principal Investigator, GEMMA V ESPÍ LÓPEZ, PhD, Principal Investigator, University of Valencia
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: ID0019
Record Dates: First submitted 2018-05-30; First posted 2018-06-21 (Actual); Last update posted 2025-07-16 (Actual); Status verified 2025-07

CONDITIONS: Low Back Pain
Keywords: low back pain; manual therapy; hypopressive therapeutic exercises
MeSH Terms: conditions — Low Back Pain | interventions — Musculoskeletal Manipulations

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Manual Therapy (Active Comparator): Manual Therapy Protocol
  1. Articulation technique L4-S1
  2. Lumbar neuromuscular technique
  3. Fascial technique of crossed hands
  4. Posteroanterior mobilizations of the lumbar vertebrae
  Interventions: Other: Manual Therapy
- Hypopressive exercises (Experimental): Protocol of 5 Hypopressive Exercises
  Interventions: Other: Hypopressive exercises

INTERVENTIONS:
Other: Manual Therapy — 1. Articulation technique L4-S1
  2. Lumbar neuromuscular technique
  3. Fascial technique of crossed hands
  4. Posteroanterior mobilizations of the lumbar vertebrae
  Arms: Manual Therapy
Other: Hypopressive exercises — Protocol 5 Hypopressive exercises
  Arms: Hypopressive exercises

SUMMARY:
Introduction Non-specific low back pain is very prevalent in our society. Different effective physiotherapy treatments have been performed in the reduction of pain and improvement of quality of life, however there are few studies that exist on the effectiveness of these treatments in protocol format based on manual therapy. On the other hand, there are no studies that implement a protocol of therapeutic exercises called abdominal hypopressives.

The aim of the study is to study the effect of a manual therapy protocol on non-specific low back pain and the implementation of hypopressive exercises in different areas such as disability, pain, flexibility and quality of life.

Material and methods

Participants The sample will consist of subjects with non-specific low back pain. Inclusion criteria

-Participants with nonspecific lumbar pain of at least 4 pain crises a month with recurrent low back pain.

Exclusion criteria

* Light acute.
* Lumbalgia after trauma.
* Presenting sciatica or musculoskeletal disorders or injuries within three months prior to the study.
* Contraindication of one of the two treatments.
* Participate in this period of no functional recovery program or physiotherapy treatment.

Study design A randomized clinical trial will be conducted. The sample will be divided into 2 groups: Group 1 will receive a manual therapy protocol that has previously shown its effectiveness in non-specific low back pain being 1 session a week, while group 2 will receive a protocol of hypopressive therapeutic exercises.

Evaluations

At the beginning of the study, a clinical interview will be carried out and, in addition, 3 evaluations will be carried out: at the beginning, at the end of the treatment and one follow-up per month. The investigators will use the following evaluation tools:

* Pain, through the Visual Analog Scale.
* Oswestry Low Back Pain Disability Scale.
* SF-36 quality of life scale.
* Visual Analog Scale.
* Algometry of spinous processes and lumbar muscles.
* Lumbar flexion with inclinometer and fingers test - floor.

ELIGIBILITY:
Inclusion Criteria:

* Man between 18 and 40 years old
* Recurrent episodes of low back pain at least 4 times a month
* At least 3 months of evolution
* Non-specific low back pain
* Not having undergone surgery

Exclusion Criteria:

* Acute low back pain
* Lumbalgia operated surgically
* Low back pain after traumatism
* Episodes of sciatica
* Contraindication to any of the treatments
* Attend, during the study period, rehabilitation programs
* Serious injuries in the 3 months prior to the study
* Root pain
* Any breach of the inclusion criteria

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 64 (Actual)
Dates: Start 2018-07-01 (Actual); Primary Completion 2018-07-31 (Actual); Study Completion 2018-09-15 (Actual)

PRIMARY OUTCOMES:
Intensity of pain | 8 weeks
  Visual Analog Scale. The participants are asked to mark the intensity of pain from 1 to 10, with 1 being almost non-existent and 10 being the worst pain imaginable.

SECONDARY OUTCOMES:
Low Back Pain Disability | 8 weeks
  Oswestry Low Back Pain Disability Scale.
  Oswestry Low Back Pain Scale: The questionnaire consists of 10 questions in which he assesses the impact of the patient's back pain on daily life activities:
  * Intensity of perceived pain
  * Personal care
  * Lift weight
  * Walk
  * Sit
  * Standing
  * Sleeping
  * Sex life
  * Social life
  * traveling There are 6 possible answers to each item being scored from 0 to 5, so that when completing the questionnaire, the scores of each item are added, multiplied by two, and we obtain a percentage over 100 of the degree of disability.
Algometry of spinous processes and lumbar muscles. | 8 weeks
  The evaluation of muscle pain was performed by algometry. The algometer evaluates the perceptual sensitivity of the pain through the pressure threshold looking for the stimulation of the nociceptors with a minimum pressure necessary to trigger discomfort at a certain point and the tolerance of the patient. The evaluator locates the point and places the pointer of the perpendicular algometer increasing the pressure force with a constant speed of 1Kg / cm² / s in a uniform and continuous way until the perception of the sensitive point, the patient informs the evaluator, he stops exerting pressure and take the corresponding record, so that the evaluator can not see the results. Between measurements, an interval of 30 seconds is left.
Lumbar flexion | 8 weeks
  Lumbar flexibility. It was measured with the Sit-and-reach (SR) test. It has been used to assess the overall flexibility on the finger-floor distance method. The test is conducted with a box designed for this purpose which has a vertical scale with a range of 50 cm (25 cm negative and 25cm positive). The subject remains standing on it, leaving the arms and trunk relaxed, then flexes the trunk forward and maintains its maximum flexion for 3 seconds. The evaluator is placed next to the scale and records the furthest measurement touched by the fingertips of both hands. If each hand reaches a different measurement, then the shortest one is registered. This is repeated 3 times and the most favourable measurement is registered.
Health status | 8 weeks
  SF-36 is a health questionnaire, both physical and metal. It contains 36 items comprising 8 health status sub-scales. It includes different dimensions (Bodily Pain, Perceptions, Mental Health, Physical Function, Role-physical, Role-emotional, Social Function, and Vitality). Positive and negative health statuses are assessed. To evaluate each dimension, the items are transformed on a scale from 0 to 100. The result is obtained by summation of all the questions, in which 0 is the worst and 100 the best result and state of health.

CONTACTS AND LOCATIONS:
Locations (1):
- Gemma v. Espí López, Valencia, Spain